CLINICAL TRIAL: NCT00824226
Title: Effect of Magnesium Treatment on Plasma Calcium in Hypoparathyroid Patients
Brief Title: Magnesium Treatment in Hypoparathyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Vallo Volke, Dr., University of Tartu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UT296
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Hypoparathyroidism
Keywords: primary hypoparathyroidism; secondary hypoparathyroidism; magnesium
MeSH Terms: conditions — Hypoparathyroidism | interventions — Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: magnesium — magnesium 350 mg tablets once a day for 3 weeks

SUMMARY:
Study hypothesis: supplementary magnesium may influence the blood calcium level in treated hypoparathyroid patients. Patients will be treated with supplementary magnesium (350 mg/day) for 3 weeks. Calcium and other relevant blood parameters will be measured before the treatment, at the end of treatment and 2 weeks after stopping treatment.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary hypoparathyroidism
* treatment with calcium plus vitamin D analogue
* ionized calcium 1,0-1,29 mmol/L
* magnesium level 0,7-1,05 mmol/L
* TSH 0.1- 10 imU/L

Exclusion Criteria:

* any other disease known to influence plasma Ca level
* pregnancy
* creatinine > 150 microM/L
* patient has used supplementary magnesium within 2 previous months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Calcium level at the end of magnesium treatment compared to pretreatment level | 3 weeks

SECONDARY OUTCOMES:
Calcium level after stopping treatment compared to the level at the end of magnesium treatment | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vallo Volke, MD, PhD, Principal Investigator — University of Tartu, Institute of Physiology
Locations (1):
- Tartu University Hospital, Tartu, Estonia